CLINICAL TRIAL: NCT04561648
Title: Standard vs High Dose of Unfractionated Heparin in the Incidence of Radial Artery Occlusion (DEFINITION) Trial.
Acronym: DEFINITION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Julio Ivan Farjat Pasos, Co-Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INCAR-DG-DI-205-2020
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Radial Artery Occlusion
Keywords: Radial Artery Occlusion; Percutaneous coronary intervention; Transradial access; Unfractionated Heparin; Coronary angiography
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: Patients that are planned to go to an invasive coronary artery angiography with good radial pulse and using the TRA are going to be randomized to two groups. One will receive the standard UFH dose and the other will receive the prespecified high dose (per Kg of body weight) of UFH.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose of Unfractionated Heparin (Experimental): 100 IU/Kg of Unfractionated Heparin
  Interventions: Drug: Unfractionated Heparin
- Standard Dose of Unfractionated Heparin (Active Comparator): 5000 IU of Unfractionated Heparin.
  Interventions: Drug: Unfractionated Heparin

INTERVENTIONS:
Drug: Unfractionated Heparin — Before removing the introducer sheath, the 2nd operator will pass the missing UFH dose to the first operator to reach 100 IU per kg of body weight in a 10 ml syringe mixed with 0.9% saline solution. The blinded first operator will administer this without knowing if it is saline or the supplemental dose of unfractionated heparin.

SUMMARY:
Double blind single center clinical trial to compare the incidence of radial artery occlusion (RAO) using standard doses of Unfractionated Heparin (UFH) vs. high doses of UFH.

DETAILED DESCRIPTION:
Radial artery occlusion (RAO) is one of the most common complications in transradial artery interventions (up to 30% of cases if specific measures are not taken to prevent it) and is related to the prothrombotic state of the patient, the scarce distal flow to the access site and the trauma caused to the artery during the procedure.

Currently worldwide, the transradial (TRA) access is the most widely used access for coronary angiography (in up to 90% of the procedures) because the transradial approach is associated with lower rates of vascular complications and event mortality (compared to the femoral access).

Although TRA access is safer, it is not free of complications, being one of the most important the RAO.

There are universal efforts to reduce RAO improving every aspects of the technique, from the type of introducer to the hemostasis time to a distal TRA, with evidence suggesting that higher doses of UFH can also decrease RAO to a greater extent. The decrease in the incidence of RAO have been proposed to be up to 2.8 times with high doses of UFH (single-center, retrospective study that compared regular not standard doses of UFH versus higher doses of UFH) although no proper prospective clinical trial have been undertaken to prove this.

The standard dose that has shown a lower rate of RAO is 5000 IU, which will be compared with 100 IU / Kg of UFH, with a randomized, prospective, double-blind design, with short-term (24-hour) follow-up with Doppler ultrasound (DUS) and its correlation with plethysmography to document RAO, and in occluded arteries, there will be a 30-day follow-up to determine the recanalization (or persistent occlusion) rates by DUS (and plethysmography). In order to address safety concerns of higher UFH doses, all the potential hemorrhagic complications will be evaluated during the study follow-up time and higher hemorrhagic risk patients are going to be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, both genders.
* Successful transradial acess for an elective diagnostic coronary angiography.

Exclusion Criteria:

* Weight <50 Kg
* Puncture of the ipsilateral radial artery in the last month.
* Still ongoing effect of pre-procedural recently used oral anticoagulants.
* Use of enoxaparin in the past in the last 12 hours prior to the procedure.
* Use of unfractionated heparin in the last 6 hours prior the procedure
* Alterations in coagulation or platelets prone to bleeding or thrombotic complications.
* Anatomical alterations at the radial access site or radial artery.
* Arteriovenous fistula in the ipsilateral arm.
* History of major bleeding associated with the use of UFH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1988 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Radial artery occlusion (RAO). | 24 hours.
  The incidence of RAO (with DUS and plethysmography).
Radial artery occlusion (RAO). | 30 days.
  The incidence of RAO (with DUS and plethysmography).

SECONDARY OUTCOMES:
Time to hemostasis. | 24 hours.
  Time to hemostasis, from the removal of the introducer sheath to hemostasis.
Diameters of the radial artery. | 24 hours.
  Minimum, maximum and mean diameters of the radial artery by vascular ultrasound.
Correlation of RAO by oximetric plethysmography and DUS. | 30 days.
  Correlation of plethysmography and DUS for the determination of RAO.
Hemorrhagic Complications. | 30 days.
  Compare the incidence of bleeding complications according to The Bleeding Academic Research Consortium 2 (BARC-2) scale:
  The BARC-2 scale:
  * Type 0
  * Type 1
  * Type 2
  * Type 3
  * Type 4
  * Type 5
Hemorrhagic Complications. | 24 hours.
  Compare the incidence of bleeding complications according to the Early Discharge After Transradial Stenting of Coronary Arteries Study (EASY) scale:
  The EASY scale:
  * Grade I
  * Grade II
  * Grade III
  * Grade IV
  * Grade V

CONTACTS AND LOCATIONS:
Overall Officials: Guering Eid Lidt, M.D., Study Director — Instituto Nacional de Cardiología Ignacio Chávez; Julio I Farjat Pasos, M.D., Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez; Carlos Aguila Bravo, M.D., Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez; Monserrat Villalobos Pedroza, M.D., Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez
Locations (1):
- Instituto Nacional de Cardiología Ignacio Chávez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No
The individual patient data will not be shared with other researchers.